CLINICAL TRIAL: NCT07162298
Title: A Randomized, Open, Single Center Clinical Study of Dragon Boat Race Versus Family Unsupervised Training to Improve the Physical Function and Quality of Life in Breast Cancer Patients
Brief Title: Dragon Boat Race Versus Family Unsupervised Training to Improve the Physical Function and Quality of Life in Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250005C
Record Dates: First submitted 2025-07-22; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Post-operation; Dragon Boat Race; Physical function; Quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dragon Boat Training Group (DB) (Experimental): The total training duration is 12 weeks, divided into cycles of 4 weeks each, with distinct training contents and goals for every cycle. Training sessions are held 3 times a week, and all participants train together on the same day. Each training session lasts approximately 60 minutes.
  In the first 4 weeks, participants spend half an hour training on land and the subsequent half an hour training on dragon boats.
  Then, from week 4 to week 8, they train for 20 minutes on land and 40 minutes on dragon boats.
  Finally, from week 8 to week 12, they only conduct 10-15 minutes of land training (as warm-up) followed by nearly an hour of on-boat training.
  This progressive training plan is designed to ensure that each participant can tolerate the training intensity as much as possible, preventing injuries caused by training.
  Interventions: Other: Dragon Boat Training
- Home-based Unsupervised Training Group (HG) (Active Comparator): The total training duration is 12 weeks. After a 15-minute warm-up (including walking, exercises, etc.), participants will perform the following 10 movements in sequence: squats, rowing simulation with rubber bands, lateral raises, sit-ups, shoulder presses, alternating bilateral lunges, dumbbell curls (for biceps), sit-ups, and planks.
  Each movement lasts 60 seconds, with a 10-second rest allowed midway through the same movement (i.e., 15 seconds of exercise followed by a 10-second rest, then another 15 seconds to complete the movement). A 20-second rest is permitted before moving on to the next movement.
  Once participants can complete 30 seconds of the same movement without needing rest or adjustment, the training intensity will be increased-progressing from one round of training (10 minutes) to two rounds (20 minutes) or even three rounds (30 minutes).
  Interventions: Other: Home-based Unsupervised Training

INTERVENTIONS:
Other: Dragon Boat Training — The total training duration is 12 weeks, divided into cycles of 4 weeks each, with distinct training contents and goals for every cycle. Training sessions are held 3 times a week, and all participants train together on the same day. Each training session lasts approximately 60 minutes.
  In the first 4 weeks, participants spend half an hour training on land and the subsequent half an hour training on dragon boats.
  Then, from week 4 to week 8, they train for 20 minutes on land and 40 minutes on dragon boats.
  Finally, from week 8 to week 12, they only conduct 10-15 minutes of land training (as warm-up) followed by nearly an hour of on-boat training.
  This progressive training plan is designed to ensure that each participant can tolerate the training intensity as much as possible, preventing injuries caused by training.
  Arms: Dragon Boat Training Group (DB)
Other: Home-based Unsupervised Training — The total training duration is 12 weeks. After a 15-minute warm-up (including walking, exercises, etc.), participants will perform the following 10 movements in sequence: squats, rowing simulation with rubber bands, lateral raises, sit-ups, shoulder presses, alternating bilateral lunges, dumbbell curls (for biceps), sit-ups, and planks.
  Each movement lasts 60 seconds, with a 10-second rest allowed midway through the same movement (i.e., 15 seconds of exercise followed by a 10-second rest, then another 15 seconds to complete the movement). A 20-second rest is permitted before moving on to the next movement.
  Once participants can complete 30 seconds of the same movement without needing rest or adjustment, the training intensity will be increased-progressing from one round of training (10 minutes) to two rounds (20 minutes) or even three rounds (30 minutes).
  Arms: Home-based Unsupervised Training Group (HG)

SUMMARY:
Investigators plans to conduct a randomized, open, single center clinical study of Dragon Boat Race versus family unsupervised training to improve the physical function and quality of life in breast cancer patients to compare the effects of organized and supervised short-term dragon boat training versus unsupervised home training on body composition, physical function, and quality of life in women after breast cancer surgery. Participants will be assigned to the following intervention protocols at a 1:1 ratio:Dragon Boat Training Group (DB): Conduct 12-week dragon boat training under the guidance of professional coaches.Home-based Unsupervised Training Group (HG): Perform exercises at home independently according to instructional videos for 12 weeks.The primary outcomes are to analyze differences in body composition, physical function, and quality of life.The secondary exploratory outcomes include stratified factors such as menopausal status and surgical methods

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-75 years;
* ECOG performance status of 0-1;
* BMI between 18.0 and 30.0;
* No prior experience with dragon boat or kayaking;
* Histologically or pathologically confirmed invasive breast cancer;
* Function levels of major organs must meet the following requirements (no blood transfusion, no use of leukocyte-elevating or platelet-elevating drugs within 2 weeks before screening):

  1. Routine blood test: absolute neutrophil count (ANC) > 1.5×10⁹/L; platelet count (PLT) > 75×10⁹/L; hemoglobin (Hb) > 90g/L; lymphocyte count ≥ 1.5×10⁹/L.
  2. Blood biochemistry: total bilirubin (TBIL) < 1.5×ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 1.5×ULN; alkaline phosphatase < 2.5×ULN; blood urea nitrogen/urea (BUN/UREA) and creatinine (Cr) < 1.5×ULN.
  3. Echocardiography: left ventricular ejection fraction (LVEF) > 55%.
  4. 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) < 470 msec. For premenopausal female patients or those not surgically sterilized: effective contraceptive methods must be used during treatment and for at least 6 months after the last dose in the study treatment.
* Voluntary participation in the study, signing of informed consent, good compliance, and willingness to cooperate with follow-up.

Exclusion Criteria:

* Stage IV breast cancer.
* Inflammatory breast cancer.
* Previous receipt of anti-tumor therapy or radiotherapy for any malignant tumor, excluding cured malignant tumors such as carcinoma in situ of the cervix, basal cell carcinoma, or squamous cell carcinoma.
* Concurrent receipt of anti-tumor therapy in other clinical trials, including but not limited to chemotherapy, endocrine therapy, biological therapy, bone-modifying agent therapy, or immune checkpoint inhibitor therapy.
* Previous regular participation in physical activity (moderate to vigorous exercise at least twice a week).
* Severe heart disease or discomfort, including but not limited to the following conditions:
* Confirmed history of heart failure or systolic dysfunction (LVEF less than 50%).
* High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate greater than 100 bpm, significant ventricular arrhythmias (e.g., ventricular tachycardia), or higher-grade atrioventricular block (i.e., Mobitz II second-degree atrioventricular block or third-degree atrioventricular block).
* Angina pectoris requiring anti-anginal medication.
* Clinically significant valvular heart disease.
* ECG showing transmural myocardial infarction.
* Poorly controlled hypertension (systolic blood pressure greater than 180 mmHg and/or diastolic blood pressure greater than 100 mmHg after drug treatment).
* Uncontrolled active infection requiring treatment; history of immunodeficiency, including positive HIV test, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.
* Patients with active chronic hepatitis B or active hepatitis C (excluding hepatitis B virus carriers, hepatitis B patients stable after drug treatment [HBV-DNA test negative or < 50 IU/ml], and cured hepatitis C patients [HCV RNA test negative]).
* Patients with any other chronic diseases (such as hypertension, diabetes, coronary heart disease, COPD, etc.).
* Patients unable to tolerate moderate to vigorous exercise.
* Pregnant or lactating female patients, female patients with childbearing potential and positive baseline pregnancy test, or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial and within 6 months after the last study medication.
* Patients with severe concomitant diseases or other comorbidities that would interfere with the planned treatment, or any other conditions deemed by the researcher to make the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2028-04-07 (Estimated)

PRIMARY OUTCOMES:
BMI (kg/m²) | 1 year
  BMI (kg/m²) weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Physical function | 1 year
  Six-minute walk test (6MWT, m)：The test is conducted in an indoor, long, straight, and flat rectangular area with a 30-meter walking route, where participants walk back and forth repeatedly. They should walk at their usual pace and rhythm as much as possible, without the need for brisk walking or jogging. The distance walked by the participants after 6 minutes is recorded. The formula reported by Enright and Sherrill, which is based on body mass index (BMI) and age, is used to compare with the 6-minute walk distance (6MWD) of normal healthy populations (for males: 6MWD (m) = 1140m - 5.61 × BMI (kg/m²) - 6.94 × age (years); for females: 6MWD (m) = 1017m - 6.24 × BMI (kg/m²) - 5.83 × age (years)).
Psychological status | 1 year
  Self-report measurement method used to assess people's acceptance of their own bodies, respect and care for their bodies, and protection of their bodies from unrealistic beauty standards. All items are rated on a 5-point scale (1 = never, 5 = always), and the total score is calculated as the average of all items, so a higher score reflects a higher level of body appreciation.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, China